CLINICAL TRIAL: NCT04727827
Title: A Prospective Interventional Trial of Pharmacogenomic-Guided Supportive Care in Hematopoietic Cell Transplantation
Brief Title: Pharmacogenomic-Guided Supportive Care in Hematopoietic Cell Transplantation
Acronym: IMPPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCI-HEM-BMT-IMPPACT-001
Record Dates: First submitted 2021-01-18; First posted 2021-01-27 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Hematopoietic Cell Transplantation; Oncology
Keywords: pharmacogenomic; precision medicine; pharmacy practice; bone marrow transplantation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This will be a prospective, pre/post interventional, single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacogenomic Testing (Experimental): A pharmacogenomic (PGx) panel will be performed to test for genetic variations in genes related to drug response.
  Interventions: Other: Pharmacogenomic-guided supportive care

INTERVENTIONS:
Other: Pharmacogenomic-guided supportive care — Patients undergoing hematopoietic stem cell transplantation will be genotyped and supportive care therapies tailored to identified drug-gene pairs and guideline recommendations

SUMMARY:
Hematopoietic cell transplantation (HCT) is the only curative treatment modality for many hematologic malignancies. Morbidity and mortality rates have declined drastically over the years, secondary to improvements in both transplant techniques and pharmacotherapies, including immunosuppressants, anti-infectives, analgesics and other supportive care medications. Despite advances in patient care, toxicities associated with HCT (e.g., graft-versus-host disease (GVHD), infection, pain, anxiety, depression, mucositis, nausea/vomiting) continue to pose challenges in patient care and have a significant impact on quality of life. (QOL). A recent study demonstrated subjects randomized to intensive supportive care had a clinically significant improvement in their QOL during hospitalization and up to 3 months post-transplant compared to those receiving standard care.

Further follow up evaluations have evaluated the impact of focused palliative care/symptom management on QOL metrics - inclusive of Edmonton Symptom Assessment surveys (ESAS). In other malignant settings, i.e. solid tumor, ESAS has been noted as an effective measure of symptoms control and the utilization of this assessment is linked to positive outcomes. The American Society of Clinical Oncology (ASCO) has designated QOL as the second most relevant metric for post-transplant patient care behind survival, making the optimization of supportive care pharmacotherapy a clinically relevant subject to investigate. Pharmacogenetics (PGx) uses an individual's genetic factors, such as single nucleotide polymorphisms (SNPs), to personalize therapy or dose selection. SNPs encode drug-metabolizing enzymes, transporters, and targets that can significantly impact drug efficacy and toxicity. With the growing complexity of both antineoplastics and supportive care, oncologists have less time to manage each subject's myriad of supportive care concerns by trial and error. Suboptimal management of symptoms compromises potential benefits from cancer therapy, disrupts clinic workflow, increases emergency room visits, and affects both patient satisfaction and reimbursement. Genetic variation is well documented across the human genome and affects a subject's response to medications regarding efficacy and toxicity. The genome is quickly becoming a pragmatic tool that can assist oncologists and other providers in optimizing supportive care for subjects with cancer.

DETAILED DESCRIPTION:
The investigators hypothesize that the implementation of a pharmacist-driven precision medicine service guided by HCT clinical pharmacists and Specialty Pharmacy pharmacists using preemptive pharmacogenomic (PGx) testing will identify drug-gene interactions relevant to the supportive care of HCT subjects. This approach to care may improve symptom management and QOL as interpreted via ESAS in adult HCT subjects treated at our institution. With the experience of past studies and a customized genetic panel, the investigators will genotype subjects prior to transplant and identify actionable drug-gene pairs and utilize these to direct supportive therapies. To date no studies have highlighted the significance of incorporating preemptive PGx testing to personalize therapy selection and dosing into the management of adult HCT subjects as a means of improving QOL and symptom management. The primary aim is to estimate the frequency of subjects undergoing PGx testing who receive at least one drug/dose selection or modification based on their test results during the study period (from admission for HCT to HCT D100). Secondarily the investigators will measure improvement in aggregate and individual scores on the ESAS survey and will further use the ESAS in its totality to assess the impact of PGx-guided care as compared to pre-implementation/non-PGx driven strategies through aggregate ESAS scores, individual ESAS scores, and differences between HCT admission (or baseline) and HCT Day 30 scores before and after the intervening program. In the outpatient setting the investigators will utilize planned medication reconciliation (with PGx guidance) by Specialty Pharmacy Service pharmacists to adhere to PGx-recommendations and capture insight into the implementation of this program to share with other practitioners. The implementation of this study will personalize pharmacotherapy, improve symptom management and QOL in adult HCT subjects treated at our institution, and offer guidance globally in supporting the role of the pharmacist in pharmacogenomics (PGx) and management of HCT subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information
* Age ≥ 18 years at the time of consent
* Scheduled HCT (allogeneic and autologous, any conditioning regimen) treatment for any malignant or non-malignant indications (i.e. aplastic anemia)
* Ability to read and understand English or Spanish
* Able to provide a buccal sample for DNA extraction and genotyping

Exclusion Criteria:

* Psychiatric illness/social situations, or active/recent (within 30 days) history of elicit substance abuse that would limit compliance with study requirements as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects undergoing PGx testing who receive at least one drug/dose selection or modification. | from admission for HCT to HCT Day +100
  The primary objective is to estimate the frequency of subjects undergoing PGx testing who receive at least one drug/dose selection or modification based on their test results during the study period

SECONDARY OUTCOMES:
Improvements in symptoms from PGx-guided supportive care | HCT admission
  Determine if PGx-guided supportive care is associated with changes in symptom management following HCT compared to control data attained from subjects not consenting to PGx testing, as assessed by individual and aggregate Edmonton Symptom Assessment Scale (ESAS) scores as well as their changes in ESAS scores (ESAS being an 11-point symptoms assessment with low scores associated with low symptom burden and the high scores associated with significant burden)
Improvements in symptoms from PGx-guided supportive care | HCT Day +30
  Determine if PGx-guided supportive care is associated with changes in symptom management following HCT compared to control data attained from subjects not consenting to PGx testing, as assessed by individual and aggregate Edmonton Symptom Assessment Scale (ESAS) scores as well as their changes in ESAS scores (ESAS being an 11-point symptoms assessment with low scores associated with low symptom burden and the high scores associated with significant burden)
Longitudinal symptoms measurements with PGx-guided supportive care | From baseline to Day +30, Day +60 and Day +100 in those who enroll to the study
  Describe longitudinal changes in individual and aggregate Edmonton Symptom Assessment Scale (ESAS) scores as indicative of QOL (ESAS being an 11-point symptoms assessment with low scores associated with low symptom burden and the high scores associated with significant burden)
Determine the type and frequency of actionable genetic polymorphisms observed in the evaluable population and in the subset that received a drug and/or dose selection/modification | From baseline to Day +30 in those who enroll to the study
  Among the PGx-guided supportive care subjects, investigators will assess the type and frequency of actionable genetic polymorphisms observed in the evaluable population and in the subset that received a drug and/or dose selection/modification based on PGx results
Determine the type and frequency of actionable genetic polymorphisms observed in the evaluable population and in the subset that received a drug and/or dose selection/modification | From baseline to Day +60 in those who enroll to the study
  Among the PGx-guided supportive care subjects, investigators will assess the type and frequency of actionable genetic polymorphisms observed in the evaluable population and in the subset that received a drug and/or dose selection/modification based on PGx results
Determine the type and frequency of actionable genetic polymorphisms observed in the evaluable population and in the subset that received a drug and/or dose selection/modification | From baseline to Day +100 in those who enroll to the study
  Among the PGx-guided supportive care subjects, investigators will assess the type and frequency of actionable genetic polymorphisms observed in the evaluable population and in the subset that received a drug and/or dose selection/modification based on PGx results

CONTACTS AND LOCATIONS:
Overall Officials: Justin R Arnall, PharmD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
All data and records generated during this study will be kept confidential in accordance with Institutional policies on subject privacy and HIPAA and that the investigator and other site personnel will not use such data and records for any purpose other than conducting the study. We do not anticipate any breach of confidentiality as no records will be shared with any personnel outside the research team. All medical information will be recorded and stored in a database. The database will exist on a password protected secured server. Medical records data will be abstracted by the Research Designee. All records will be kept confidential.

REFERENCES:
- [Background] Sureda A, Bader P, Cesaro S, Dreger P, Duarte RF, Dufour C, Falkenburg JH, Farge-Bancel D, Gennery A, Kroger N, Lanza F, Marsh JC, Nagler A, Peters C, Velardi A, Mohty M, Madrigal A. Indications for allo- and auto-SCT for haematological diseases, solid tumours and immune disorders: current practice in Europe, 2015. Bone Marrow Transplant. 2015 Aug;50(8):1037-56. doi: 10.1038/bmt.2015.6. Epub 2015 Mar 23. PMID 25798672
- [Background] El-Jawahri A, LeBlanc T, VanDusen H, Traeger L, Greer JA, Pirl WF, Jackson VA, Telles J, Rhodes A, Spitzer TR, McAfee S, Chen YA, Lee SS, Temel JS. Effect of Inpatient Palliative Care on Quality of Life 2 Weeks After Hematopoietic Stem Cell Transplantation: A Randomized Clinical Trial. JAMA. 2016 Nov 22;316(20):2094-2103. doi: 10.1001/jama.2016.16786. PMID 27893130
- [Background] McCabe MS, Bhatia S, Oeffinger KC, Reaman GH, Tyne C, Wollins DS, Hudson MM. American Society of Clinical Oncology statement: achieving high-quality cancer survivorship care. J Clin Oncol. 2013 Feb 10;31(5):631-40. doi: 10.1200/JCO.2012.46.6854. Epub 2013 Jan 7. No abstract available. PMID 23295805
- [Background] Evans WE, McLeod HL. Pharmacogenomics--drug disposition, drug targets, and side effects. N Engl J Med. 2003 Feb 6;348(6):538-49. doi: 10.1056/NEJMra020526. No abstract available. PMID 12571262
- [Background] Patel JN, Wiebe LA, Dunnenberger HM, McLeod HL. Value of Supportive Care Pharmacogenomics in Oncology Practice. Oncologist. 2018 Aug;23(8):956-964. doi: 10.1634/theoncologist.2017-0599. Epub 2018 Apr 5. PMID 29622698
- [Background] Owusu Obeng A, Hamadeh I, Smith M. Review of Opioid Pharmacogenetics and Considerations for Pain Management. Pharmacotherapy. 2017 Sep;37(9):1105-1121. doi: 10.1002/phar.1986. Epub 2017 Sep 6. PMID 28699646
- [Background] Ciszkowski C, Madadi P, Phillips MS, Lauwers AE, Koren G. Codeine, ultrarapid-metabolism genotype, and postoperative death. N Engl J Med. 2009 Aug 20;361(8):827-8. doi: 10.1056/NEJMc0904266. No abstract available. PMID 19692698
- [Background] Crews KR, Gaedigk A, Dunnenberger HM, Leeder JS, Klein TE, Caudle KE, Haidar CE, Shen DD, Callaghan JT, Sadhasivam S, Prows CA, Kharasch ED, Skaar TC; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium guidelines for cytochrome P450 2D6 genotype and codeine therapy: 2014 update. Clin Pharmacol Ther. 2014 Apr;95(4):376-82. doi: 10.1038/clpt.2013.254. Epub 2014 Jan 23. PMID 24458010
- [Background] Hicks JK, Bishop JR, Sangkuhl K, Muller DJ, Ji Y, Leckband SG, Leeder JS, Graham RL, Chiulli DL, LLerena A, Skaar TC, Scott SA, Stingl JC, Klein TE, Caudle KE, Gaedigk A; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for CYP2D6 and CYP2C19 Genotypes and Dosing of Selective Serotonin Reuptake Inhibitors. Clin Pharmacol Ther. 2015 Aug;98(2):127-34. doi: 10.1002/cpt.147. Epub 2015 Jun 29. PMID 25974703
- [Background] Altar CA, Carhart J, Allen JD, Hall-Flavin D, Winner J, Dechairo B. Clinical Utility of Combinatorial Pharmacogenomics-Guided Antidepressant Therapy: Evidence from Three Clinical Studies. Mol Neuropsychiatry. 2015 Oct;1(3):145-55. doi: 10.1159/000430915. Epub 2015 Jul 31. PMID 27606312
- [Background] Perez V, Salavert A, Espadaler J, Tuson M, Saiz-Ruiz J, Saez-Navarro C, Bobes J, Baca-Garcia E, Vieta E, Olivares JM, Rodriguez-Jimenez R, Villagran JM, Gascon J, Canete-Crespillo J, Sole M, Saiz PA, Ibanez A, de Diego-Adelino J; AB-GEN Collaborative Group; Menchon JM. Efficacy of prospective pharmacogenetic testing in the treatment of major depressive disorder: results of a randomized, double-blind clinical trial. BMC Psychiatry. 2017 Jul 14;17(1):250. doi: 10.1186/s12888-017-1412-1. PMID 28705252
- [Background] Winner JG, Carhart JM, Altar CA, Allen JD, Dechairo BM. A prospective, randomized, double-blind study assessing the clinical impact of integrated pharmacogenomic testing for major depressive disorder. Discov Med. 2013 Nov;16(89):219-27. PMID 24229738
- [Background] Nassan M, Nicholson WT, Elliott MA, Rohrer Vitek CR, Black JL, Frye MA. Pharmacokinetic Pharmacogenetic Prescribing Guidelines for Antidepressants: A Template for Psychiatric Precision Medicine. Mayo Clin Proc. 2016 Jul;91(7):897-907. doi: 10.1016/j.mayocp.2016.02.023. Epub 2016 Jun 21. PMID 27289413
- [Background] Bousman CA, Forbes M, Jayaram M, Eyre H, Reynolds CF, Berk M, Hopwood M, Ng C. Antidepressant prescribing in the precision medicine era: a prescriber's primer on pharmacogenetic tools. BMC Psychiatry. 2017 Feb 8;17(1):60. doi: 10.1186/s12888-017-1230-5. PMID 28178974
- [Background] Trammel M, Roederer M, Patel J, McLeod H. Does pharmacogenomics account for variability in control of acute chemotherapy-induced nausea and vomiting with 5-hydroxytryptamine type 3 receptor antagonists? Curr Oncol Rep. 2013 Jun;15(3):276-85. doi: 10.1007/s11912-013-0312-x. PMID 23512709
- [Background] Chen JS, Li LS, Cheng DR, Ji SM, Sun QQ, Cheng Z, Wen JQ, Sha GZ, Liu ZH. Effect of CYP3A5 genotype on renal allograft recipients treated with tacrolimus. Transplant Proc. 2009 Jun;41(5):1557-61. doi: 10.1016/j.transproceed.2009.01.097. PMID 19545678
- [Background] Quteineh L, Verstuyft C, Furlan V, Durrbach A, Letierce A, Ferlicot S, Taburet AM, Charpentier B, Becquemont L. Influence of CYP3A5 genetic polymorphism on tacrolimus daily dose requirements and acute rejection in renal graft recipients. Basic Clin Pharmacol Toxicol. 2008 Dec;103(6):546-52. doi: 10.1111/j.1742-7843.2008.00327.x. PMID 19067682
- [Background] Tang HL, Xie HG, Yao Y, Hu YF. Lower tacrolimus daily dose requirements and acute rejection rates in the CYP3A5 nonexpressers than expressers. Pharmacogenet Genomics. 2011 Nov;21(11):713-20. doi: 10.1097/FPC.0b013e32834a48ca. PMID 21886016
- [Background] Abidi MZ, D'Souza A, Kuppalli K, Ledeboer N, Hari P. CYP2C19*17 genetic polymorphism--an uncommon cause of voriconazole treatment failure. Diagn Microbiol Infect Dis. 2015 Sep;83(1):46-8. doi: 10.1016/j.diagmicrobio.2015.05.002. Epub 2015 May 7. PMID 25986028
- [Background] Bennis Y, Bodeau S, Bouquie R, Deslandes G, Verstuyft C, Gruson B, Andrejak M, Lemaire-Hurtel AS, Chouaki T. High metabolic N-oxidation of voriconazole in a patient with refractory aspergillosis and CYP2C19*17/*17 genotype. Br J Clin Pharmacol. 2015 Oct;80(4):782-4. doi: 10.1111/bcp.12713. Epub 2015 Aug 24. No abstract available. PMID 26138512
- [Background] Cendejas-Bueno E, Borobia AM, Gomez-Lopez A, Escosa-Garcia L, Rio-Garcia M, Plaza D, Garcia-Rodriguez J, Carcas-Sansuan A. Invasive aspergillosis in a paediatric allogeneic stem cell transplantation recipient owing to a susceptible Aspergillus fumigatus: Treatment failure with high doses of voriconazole and influence of CYP2C19 polymorphisms. Int J Antimicrob Agents. 2016 May;47(5):410-1. doi: 10.1016/j.ijantimicag.2016.02.002. Epub 2016 Feb 27. No abstract available. PMID 27056297
- [Background] Moriyama B, Jarosinski PF, Figg WD, Henning SA, Danner RL, Penzak SR, Wayne AS, Walsh TJ. Pharmacokinetics of intravenous voriconazole in obese patients: implications of CYP2C19 homozygous poor metabolizer genotype. Pharmacotherapy. 2013 Mar;33(3):e19-22. doi: 10.1002/phar.1192. Epub 2013 Feb 11. PMID 23400848
- [Background] Moriyama B, Falade-Nwulia O, Leung J, Penzak SR, JJingo C, Huang X, Henning SA, Wilson WH, Walsh TJ. Prolonged half-life of voriconazole in a CYP2C19 homozygous poor metabolizer receiving vincristine chemotherapy: avoiding a serious adverse drug interaction. Mycoses. 2011 Nov;54(6):e877-9. doi: 10.1111/j.1439-0507.2011.02016.x. Epub 2011 May 25. PMID 21615537
- [Background] Andersen RL, Johnson DJ, Patel JN. Personalizing supportive care in oncology patients using pharmacogenetic-driven treatment pathways. Pharmacogenomics. 2016 Mar;17(4):417-34. doi: 10.2217/pgs.15.178. Epub 2016 Feb 12. PMID 26871520
- [Background] Patel JN, Robinson MM, Hamadeh I, et al: CYP2C19 Genotype-Guided Dosing and Voriconazole Concentrations in Hematopoietic Stem Cell Transplant Patients (HSCT) Receiving Antifungal Prophylaxis. Blood 128, 2016; abstr 3416
- [Background] Crews KR, Cross SJ, McCormick JN, Baker DK, Molinelli AR, Mullins R, Relling MV, Hoffman JM. Development and implementation of a pharmacist-managed clinical pharmacogenetics service. Am J Health Syst Pharm. 2011 Jan 15;68(2):143-50. doi: 10.2146/ajhp100113. PMID 21200062
- [Background] Dunnenberger HM, Crews KR, Hoffman JM, Caudle KE, Broeckel U, Howard SC, Hunkler RJ, Klein TE, Evans WE, Relling MV. Preemptive clinical pharmacogenetics implementation: current programs in five US medical centers. Annu Rev Pharmacol Toxicol. 2015;55:89-106. doi: 10.1146/annurev-pharmtox-010814-124835. Epub 2014 Oct 2. PMID 25292429

DOCUMENTS (1):
  • Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04727827/ICF_000.pdf